CLINICAL TRIAL: NCT05859620
Title: Implementation of a Clinical Screening and Response System for the Early Detection of Cardiac Complications After Noncardiac Surgery: Feasibility and Medicoeconomic Impact
Brief Title: Implementation of a Clinical Screening and Response System for Cardiac Complications After Noncardiac Surgery
Acronym: ImplementPMI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Luzerner Kantonsspital (Other); Kantonsspital Olten (Other); Medical University Innsbruck (Other); University Hospital, Geneva (Other); Bürgerspital Solothurn (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02899
Record Dates: First submitted 2023-02-06; First posted 2023-05-16 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Myocardial Injury; Myocardial Infarction; Perioperative Complication
Keywords: Myocardial injury; Myocardial infarction; Perioperative care; Noncardiac surgery; Screening
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before implementation: Patients included before implementation of the PMI-screening
  Interventions: Other: Patient assessment and follow-up
- After implementation: Patients included after implementation of the PMI-screening
  Interventions: Other: Patient assessment and follow-up

INTERVENTIONS:
Other: Patient assessment and follow-up — There is no study-specific intervention. The investigators will record data generated by clinical activity before, during and after implementation of the PMI-screening. Follow-up data and the final PMI event adjudication will be the only data generated specifically for this study.

SUMMARY:
The investigators aim to show the feasibility and medicoeconomic impact of implementing a clinical screening and response system for the early detection of perioperative cardiac complications in high-risk patients.

Specifically, the investigators aim to: 1) evaluate the feasibility of implementation of a PMI-screening; 2) evaluate the medicoeconomic impact of implementing a PMI-screening; 3) identify barriers to implementation; 4) generate data for a future randomized controlled trial on outcomes by exploring opportunities to improve care following PMI, the occurrence and timing of major adverse cardiac events (MACE), and the treatment effect associated with PMI-screening.

DETAILED DESCRIPTION:
Background: Perioperative myocardial infarction/injury (PMI) is increasingly recognised as frequent, but often undiagnosed and untreated contributor to mortality following noncardiac surgery. Due to differences in pathophysiology and perioperative anaesthesia and analgesia, most PMI do not cause typical ischemic symptoms and are therefore missed in routine clinical practice. Active surveillance using cardiac troponin (cTn) is now guideline-recommended for the early detection of PMI to possibly improve outcome1. Given substantial concerns regarding the feasibility and health economic impact of implementing such a strategy, it is not yet widely applied.

Aim: to show feasibility of implementation as well as health economic impact of an active surveillance for the early detection of PMI in high-risk patients.

Methodology: in this observational before-after study the investigators will enrol patients at high cardiovascular risk undergoing noncardiac surgery before and after implementation of a PMI screening. Patients in the pre-implementation phase will receive standard of care, while in the post-implementation phase patients receive a PMI-screening, consisting of a preoperative and two postoperative measurements of high-sensitivity cTn (hs-cTn) and a cardiology consultation will be done in case of detection of a PMI. Patient data, resource utilisation, and PMI-aetiology will be collected. Interviews with key stakeholders will identify barriers to implementation. One-year follow-up will be conducted to evaluate occurrence of death, MACE, and safety endpoints.

Potential significance: This study will generate important insights regarding the feasibility, safety and the health economic impact of implementing an active surveillance for the early detection of PMI.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients fulfilling the institutional criteria for inclusion into the routine PMI-screening
* aged 40-85 years
* at increased cardiovascular risk
* undergoing inpatient, noncardiac, elective or emergent surgery
* postoperative stay of ≥2 nights at the participating institution
* orthopaedic, traumatology, vascular, spinal, thoracic, neurosurgical, and visceral surgery.

Exclusion Criteria:

* patients with cardiac surgery or interventions in the last 14 days
* chronic renal failure under dialysis, renal transplant surgery
* moderate-to-severe dementia
* previous inclusion within 5 days
* documented refusal to use of their data for research purposes or refusal of further use during follow-up
* Patients declining consent for follow-up will be excluded from follow-up analyses.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 40-85 years at increased cardiovascular risk undergoing inpatient, noncardiac, elective or emergent surgery with a planned postoperative stay of ≥2 nights
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Perioperative Myocardial Infarction/Injury (PMI)-Screening (Reach) | during the hospital stay (up to postoperative day 2)
  Percentage of patients eligible for PMI-screening according to inclusion criteria, but not screened during the implementation phase (defined as no or only one measurement of hs-cTn done during screening days)
Incidence of PMI | after the surgery until postoperative day 2
  Percentage of patients experiencing PMI following noncardiac surgery
Cardiology consultation (Fidelity) | during hospital stay (up to postoperative day 5)
  Percentage of patients with detected PMI by PMI-screening on screening days, seen vs. not seen by a cardiologist
Diagnostic challenge | during hospital stay (up to postoperative day 5)
  Number of cases with mismatch of initial classification of PMI aetiology (and management pathway) at time of consultation versus final adjudication. In case of two differential diagnoses stated on the cardiology consultation, mismatch is seen when none of the diagnoses correspond to the final adjudication. If three or more differential diagnoses are stated, mismatch is seen in any case even if the final adjudication diagnosis is stated
Barriers to implementation | following the post-implementation period (6 months after implementation)
  Barriers to implementation will be assessed by a semi-quantitive questionnaire complemented by qualitative focus group including the local investigators and representatives of cardiology and anaesthesiology

SECONDARY OUTCOMES:
Medicoeconomic impact | Within 3 - 30 days following surgery
  Cost of postoperative blood draws on day 1 and 2, length of hospital stay, days on intensive care unit, consultations within day 1-3, ECG within day 1-3, cardiac stress testing within 30 days, and cardiac catheterisation within 30 days, denoted in Swiss Francs
Resource Usage | Within 3 - 30 days following surgery
  Number of postoperative blood draws on day 1 and 2, length of hospital stay, days on intensive care unit, consultations within day 1-3, ECG within day 1-3, cardiac stress testing within 30 days, and cardiac catheterisation within 30 days
Major adverse cardiac events (MACE) | 1 year
  Occurrence and timing of a composite of major adverse cardiac events (MACE) within twelve months, consisting of: All-cause death, acute myocardial infarction Type 1, survived sudden cardiac death, and Acute heart failure
Complications of cardiology diagnostics | 30 days
  Number of inappropriate interventions or complications of cardiology diagnostics and interventions, consisting of: Overtreatment (Coronary angiographies showing normal coronaries), complications of cardiac interventions (myocardial infarction, stroke, death)
Major bleeding | Postoperative day 1 - 1 year (blinding of first 24h following surgery)
  Bleeding Academic Research Consortium Typ 3-5

CONTACTS AND LOCATIONS:
Overall Officials: Christian Puelacher, MD-PhD, Principal Investigator — University Hospital, Basel, Switzerland; Christian Müller, Prof., Study Director — University Hospital, Basel, Switzerland
Locations (5):
- University Hospital Innsbruck, Innsbruck, Tyrol, Austria
- Switzerland (4):
  - University Hospital Geneva, Geneva, Canton of Geneva
  - Cantonal Hospital Lucerne, Lucerne, Canton of Lucerne
  - Canton Hospital Olten, Olten, Canton of Solothurn
  - Bürgerspital Solothurn, Solothurn

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing with other research groups will be the responsibility of the PI.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT05859620/Prot_SAP_000.pdf